CLINICAL TRIAL: NCT02795936
Title: Feasibility of Cardiac Rehabilitation in Patients With Heart Failure at the Moi Teaching and Referral Hospital
Acronym: FCR-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Moi Teaching and Referral Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00071928
Record Dates: First submitted 2016-05-31; First posted 2016-06-10 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure
Keywords: rehabilitation; exercise
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Cardiac Rehabilitation; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Institutional based rehabilitation (Active Comparator): Conduct cardiac rehabilitation exercise protocol within the hospital
  Interventions: Procedure: Cardiac rehabilitation
- Home based rehabilitation (Active Comparator): Conduct cardiac rehabilitation exercise protocol at home
  Interventions: Procedure: Cardiac rehabilitation
- Observational arm (Placebo Comparator): No prescribed exercises, followed up monthly
  Interventions: Procedure: Cardiac rehabilitation

INTERVENTIONS:
Procedure: Cardiac rehabilitation — Perform exercise prescription for 12 weeks
  Other Names: exercise

SUMMARY:
This is a study to find out whether cardiac rehabilitation is feasible in Western Kenya.

This study will test whether cardiac rehabilitation is feasible by measuring how many participants are able to follow and complete two different exercise protocols; one at home and one in hospital. It will also measure how the exercise intervention affects quality of living, depression and improvement in exercise tolerance.

DETAILED DESCRIPTION:
Cardiovascular diseases are major drivers of global disease burden. Heart failure, has a 50% mortality at 5 years and is thought to be higher in resource limited settings. Cardiac rehabilitation (CR) is a multi-disciplinary intervention which has been demonstrated to improve functional status, quality of life, and reduce morbidity and mortality in patients with heart failure. In sub-Saharan Africa, despite a significant heart failure disease burden, CR is largely non-existent. There is a compelling need for urgent development of access to CR in the region. However, feasibility and potential utilization of CR is unknown. The investigators aim to conduct a mixed methods study to evaluate feasibility of home based and institution based CR.

Participants will be voluntarily recruited from a convenience sample at the Moi Teaching and Referral Hospital (MTRH) outpatient cardiology clinic. Based on a reasonable estimate of expected subject recruitment over the time frame of study, 25 patients will be recruited into the institution based cardiac rehabilitation (IBCR) arm. In consideration of the potentially larger population and a wider geographical spread of home based cardiac rehabilitation (HBCR), 36 patients will be recruited to the HBCR arm and 40 patients will be recruited into an observational arm. While the study is not designed to make comparative outcome inferences between the HBCR and the IBCR groups, the sample size will be large enough to detect a clinically significant mean post intervention increase in 6 minute walk time distance in the HBCR arm of 50m.

The participants will be involved in physical exercises, nutritional counseling and educational sessions. Upon completion of the rehabilitation protocols, patients from both study arms will also be invited to participate in focus group discussions. Data will be analyzed and numeric data will be expressed as number (percent), means (standard deviation) or median (interquartile range). Wilcoxon rank-sum and Fisher's exact tests for pre - post intervention comparisons of continuous and binary variables, respectively. Focus group discussions will be transcribed and analyzed to identify discussion themes.

ELIGIBILITY:
Inclusion Criteria:

1. New York Heart Association (NYHA) Class II and III heart failure
2. Have had an echocardiographic study in the past 5 years
3. Owns a mobile telephone
4. Can participate in exercise
5. Can read/ primary care giver can read in English or Kiswahili
6. Can travel to hospital three times a week

Exclusion Criteria:

1. Recent acute illness requiring hospitalization or initiation of new medication in the preceding 4 weeks
2. Limitation of activity because of factors other than fatigue or exertional dyspnea, such as arthritis, claudication in the legs, angina, advanced comorbidities
3. Known arrhythmia
4. Heart failure due to congenital heart disease
5. Pregnant patients as may be confirmed by patient report or urine pregnancy tests
6. Heart failure due to obstructive cardiomyopathy including mitral stenosis and aortic stenosis
7. Presence of implanted pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Protocol adherence | 12 weeks
  Mean adherence of at least 25% to the exercise prescriptions

SECONDARY OUTCOMES:
Change in 6 minute walk time distance (in meters) | baseline, 12 weeks
  Measure of functional capacity
Change in Depression screen score using patient health questionnaire 9 (PHQ9) | baseline, 12 weeks
  Screen score based on patient health questionnaire 9 (PHQ9)
Change in Quality of life using short form health survey (SF 36) score | baseline, 12 weeks
  Quality of life based on short form health survey (SF 36) score
Qualitative assessment of perceptions towards cardiac rehabilitation from focus group discussions | 12 weeks
  Thematic analysis of barriers and incentives towards cardiac rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Gerald S Bloomfield, MD, Principal Investigator — Duke Universisty
Locations (1):
- Moi teaching and Referral Hospital, Eldoret, Uasin Gishu County, Kenya

REFERENCES:
- [Background] Moran A, Forouzanfar M, Sampson U, Chugh S, Feigin V, Mensah G. The epidemiology of cardiovascular diseases in sub-Saharan Africa: the Global Burden of Diseases, Injuries and Risk Factors 2010 Study. Prog Cardiovasc Dis. 2013 Nov-Dec;56(3):234-9. doi: 10.1016/j.pcad.2013.09.019. Epub 2013 Sep 28. PMID 24267430
- [Background] Arroll B, Doughty R, Andersen V. Investigation and management of congestive heart failure. BMJ. 2010 Jul 14;341:c3657. doi: 10.1136/bmj.c3657. No abstract available. PMID 20630951
- [Background] Kwan G, Balady GJ. Cardiac rehabilitation 2012: advancing the field through emerging science. Circulation. 2012 Feb 21;125(7):e369-73. doi: 10.1161/CIRCULATIONAHA.112.093310. No abstract available. PMID 22354982
- [Background] Clark RA, Conway A, Poulsen V, Keech W, Tirimacco R, Tideman P. Alternative models of cardiac rehabilitation: a systematic review. Eur J Prev Cardiol. 2015 Jan;22(1):35-74. doi: 10.1177/2047487313501093. Epub 2013 Aug 13. PMID 23943649
- [Background] Binanay CA, Akwanalo CO, Aruasa W, Barasa FA, Corey GR, Crowe S, Esamai F, Einterz R, Foster MC, Gardner A, Kibosia J, Kimaiyo S, Koech M, Korir B, Lawrence JE, Lukas S, Manji I, Maritim P, Ogaro F, Park P, Pastakia SD, Sugut W, Vedanthan R, Yanoh R, Velazquez EJ, Bloomfield GS. Building Sustainable Capacity for Cardiovascular Care at a Public Hospital in Western Kenya. J Am Coll Cardiol. 2015 Dec 8;66(22):2550-60. doi: 10.1016/j.jacc.2015.09.086. PMID 26653630
- [Background] Turk-Adawi K, Sarrafzadegan N, Grace SL. Global availability of cardiac rehabilitation. Nat Rev Cardiol. 2014 Oct;11(10):586-96. doi: 10.1038/nrcardio.2014.98. Epub 2014 Jul 15. PMID 25027487
- [Derived] Ngeno GTK, Barasa F, Kamano J, Kwobah E, Wambui C, Binanay C, Egger JR, Kussin PS, Thielman NM, Bloomfield GS. Feasibility of Cardiac Rehabilitation Models in Kenya. Ann Glob Health. 2022 Jan 18;88(1):7. doi: 10.5334/aogh.3392. eCollection 2022. PMID 35087707

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT02795936/Prot_SAP_001.pdf